CLINICAL TRIAL: NCT03148236
Title: Pilot Study of the Safety and Efficacy of Intravenous Vitamin C in Patients Undergoing Atrial Fibrillation Ablation
Brief Title: Vitamin C in Atrial Fibrillation Ablation
Acronym: VitC-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20006786
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation Ablation
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Active Comparator)
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin C — 200mg/kg/day split into 4 doses infused every six hours over 30 minutes in 50ml D5W
  Other Names: Ascorbic Acid
  Arms: Vitamin C
Other: Placebo — 50mL infused over 30 minutes
  Other Names: D5W
  Arms: Placebo

SUMMARY:
Single-center, double-blinded, randomized, controlled safety and feasibility pilot study of high dose IV ascorbic acid (200mg/kg) over 24 hours, divided into four doses and administered every six hours with a 30 minute IV infusion time per dose, compared to matched placebo infusion

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 21 years
2. Diagnosis of atrial fibrillation with plans for a catheter-based ablation procedure
3. Ability to provide informed consent and willingness to be included in the study

Exclusion Criteria:

1. Known allergy to Vitamin C
2. Inability to obtain informed consent
3. Diabetes mellitus either requiring the use of insulin therapy or not requiring the use of insulin therapy but which is uncontrolled, defined as a glycosylated hemoglobin of greater than or equal to 8%
4. Prior catheter-based ablation for atrial fibrillation
5. Pregnancy or breast feeding
6. Active renal calculus
7. Active acute or chronic infection (including HIV or hepatitis C)
8. Active or recent (within 5 years) malignancy
9. Autoimmune or autoinflammatory disease
10. Recent or active use of immunosuppressive medications
11. Non-English speaking
12. Ward of the state (inmate, other)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayanthe Koneru, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trankle CR, Puckett L, Swift-Scanlan T, DeWilde C, Priday A, Sculthorpe R, Ellenbogen KA, Fowler A, Koneru JN. Vitamin C Intravenous Treatment In the Setting of Atrial Fibrillation Ablation: Results From the Randomized, Double-Blinded, Placebo-Controlled CITRIS-AF Pilot Study. J Am Heart Assoc. 2020 Feb 4;9(3):e014213. doi: 10.1161/JAHA.119.014213. Epub 2020 Jan 30. PMID 32013700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin C | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin C | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 3 | 5 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [56 to 69] | 65 [54 to 70] | 63 [56 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Creatinine Levels
Description: Change in Kidney Function
Time Frame: Baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 10 | 10
mg/dL | -0.1 [-0.2 to -0.1] | -0.1 [-0.2 to 0]

2. Primary Outcome: Change in Plasma Levels of Ascorbic Acid
Description: Change in plasma levels of ascorbic acid
Time Frame: baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 10 | 10
micromolar | 267 [98 to 597] | -4 [-8 to -1]

3. Primary Outcome: Change in hsCRP
Description: Biomarker of inflammation
Time Frame: baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 10 | 10
mg/L | 5.31 [4.48 to 7.92] | 16.01 [9.40 to 29.29]

4. Primary Outcome: Change in Interleukin (IL-6)
Description: Biomarker of inflammation
Time Frame: baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
pg/mL | 13.3 [6.6 to 29.4] | 6.6 [2.6 to 12.1]

5. Primary Outcome: Change in Von Willebrand Factor (vWF)
Description: Biomarker of blood vessel damage
Time Frame: baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: micrograms/mL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
micrograms/mL | 0.4 [-1.3 to 4.8] | 0.4 [-2.5 to 2.5]

6. Primary Outcome: Change in Creatinine Levels
Description: Change in kidney function
Time Frame: Baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
mg/dL | 0 [-0.1 to 0] | 0.1 [0 to 0.1]

7. Primary Outcome: Change in Plasma Ascorbic Acid Level
Description: Change in plasma ascorbic acid level
Time Frame: Baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
micromolar | 3 [-10 to 21] | -5 [-12 to 20]

8. Primary Outcome: Change in hsCRP
Description: Biomarker of inflammation
Time Frame: baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
mg/L | -0.30 [-1.16 to 0.32] | -0.64 [-2.70 to -0.15]

9. Primary Outcome: Change in Interleukin (IL-6)
Description: Biomarker of inflammation
Time Frame: baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
pg/mL | 0 [-0.7 to 0.4] | 0.1 [-0.6 to 1.1]

10. Primary Outcome: Change in Von Willebrand Factor (vWF)
Description: Biomarker of blood vessel damage
Time Frame: baseline to 30 days
Measure: Median (Inter-Quartile Range); unit: micrograms/mL
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 9 | 10
micrograms/mL | -2.3 [-3.7 to 1.7] | -3.8 [-7.5 to 0.6]

11. Secondary Outcome: Post Procedural Pain
Description: Sum of pain scores every six hours for the 24 hour period following ablation measured on a visual analog scale scored on a level from zero (no pain) to 10 (maximum pain)
Time Frame: baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin C | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 4.5 [1.3 to 9.8] | 0.3 [0 to 1]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Vitamin C | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C (N=10) | Placebo (N=10)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) — Pericarditis within 24 hours of the ablation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03148236/Prot_000.pdf